CLINICAL TRIAL: NCT02581345
Title: A Phase 3 Randomized, Double-blind, Multicenter Study to Evaluate Efficacy, Safety, and Immunogenicity of an Adalimumab Biosimilar (M923) and Humira® in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis
Brief Title: Phase 3 Study of M923 and Humira® in Subjects With Chronic Plaque-type Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Momenta Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 911401
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Chronic Plaque Psoriasis; Psoriasis
Keywords: Moderate to severe chronic plaque psoriasis; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- M923 (Experimental): Participants assigned to receive M923
  Interventions: Biological: M923
- Humira (Active Comparator): Participants assigned to receive Humira
  Interventions: Biological: Humira
- M923 and Humira (Other): Participants assigned to receive M923 and Humira
  Interventions: Biological: M923; Biological: Humira

INTERVENTIONS:
Biological: M923 — Recombinant human immunoglobulin G subclass 1 (IgG1) monoclonal antibody specific for human tumor necrosis factor-alpha (TNF-α)
  Other Names: Adalimumab
  Arms: M923; M923 and Humira
Biological: Humira — Recombinant human immunoglobulin G subclass 1 (IgG1) monoclonal antibody specific for human tumor necrosis factor-alpha (TNF-α)
  Other Names: Adalimumab
  Arms: Humira; M923 and Humira

SUMMARY:
The purpose of the study is to evaluate efficacy, safety, and immunogenicity of a proposed adalimumab biosimilar (M923) and Humira in participants with moderate to severe chronic plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and communicate with the investigator and comply with the requirements of the study
2. Chronic plaque-type psoriasis diagnosed for at least 6 months before screening
3. Stable plaque psoriasis
4. History of receipt of or candidate for therapy.
5. Moderate to severe psoriasis at screening and baseline
6. Must be willing and able to self-administer SC injections or have a caregiver available to administer injections
7. Male participants of childbearing potential must employ a highly effective contraceptive measure
8. Female participants must have a negative pregnancy test; are not planning to become pregnant; and must not be lactating. Female participants must also agree to employ a highly effective contraceptive measure.

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type
2. Drug-induced psoriasis.
3. Other skin conditions which would interfere with assessment of psoriasis
4. Medical conditions other than psoriasis for which systemic corticosteroids were used in the last year prior to screening
5. Other inflammatory conditions other than psoriasis or psoriatic arthritis
6. Prior use of systemic tumor necrosis factor (TNF) inhibitors, or 2 or more non-TNF biologic therapies
7. Ongoing use of prohibited psoriasis treatments
8. Ongoing use of other non-psoriasis prohibited treatments
9. All other prior non-psoriasis concomitant treatments must be on a stable dose for at least 4 weeks
10. Laboratory abnormalities at screening deemed clinically significant by the investigator
11. Any condition or illness which in the opinion of the investigator or sponsor poses an unacceptable safety risk
12. History of latex allergy
13. History of or current signs or symptoms or diagnosis of a demyelinating disorder
14. History of or current Class III or IV New York Heart Association congestive heart failure
15. Signs, symptoms, or diagnosis of lymphoproliferative disorders, lymphoma, leukemia, myeloproliferative disorders, or multiple myeloma
16. Current malignancy or history of any malignancy except adequately treated or excised non metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ; no more than 3 lifetime basal cell and squamous cell carcinomas permitted
17. Chronic infections, recurrent infections; recent infection to be evaluated
18. History of or presence of human immunodeficiency virus (HIV), or Hepatitis B (HBV) or C virus (HCV)
19. History of active tuberculosis (TB) or untreated or inadequately treated latent TB.
20. Exposure to an investigational product ≤30 days prior to enrollment or participation in another clinical study during the course of this study
21. Participant is a family member or employee of the investigator or site staff or study team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2015-09; Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Caminis, MD, Study Director — Shire
Locations (89):
- United States (24):
  - Wallace Medical Group, Inc., Beverly Hills, California
  - Encino Research Center, Encino, California
  - eStudySite, La Mesa, California
  - eStudySite, Oceanside, California
  - eStudySite, San Diego, California
  - Shahram Jacobs MD, INC, Sherman Oaks, California
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Bioclinical Research Alliance; Inc, Miami, Florida
  - Sanitas Reasearch, LLC, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, LLC, Orlando, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Radiant Research; Inc., Overland Park, Kansas
  - Tufts Medical Center; Inc., Boston, Massachusetts
  - Bay State Clinical Trials, Inc, Watertown, Massachusetts
  - eStudySite, Las Vegas, Nevada
  - Radiant Research; Inc., Cincinnati, Ohio
  - Radiant Research, Inc., Columbus, Ohio
  - Radiant Clinical Research, Anderson, South Carolina
  - Palmetto Clinical Trial Services, LLC, Fountain Inn, South Carolina
  - Radiant Research, Inc., Greer, South Carolina
  - Austin Institute for Clinical Research, LLC, Pflugerville, Texas
  - Clinical Trials of Texas; Inc., San Antonio, Texas
  - National Clinical Research-Richmond, Inc, Richmond, Virginia
- Bulgaria (5):
  - Medical Centre Asklepii, OOD, Dupnitsa
  - DCC Sveti Georgi EOOD, Haskovo
  - UMHAT Dr.Georgi Stranski, EAD, Pleven
  - DCC Sv. Georgi, EOOD, Plovdiv
  - Department of Dermatology and Venereology, Faculty of Medicine, UMHAT Alexandrovska, Sofia
- Canada (10):
  - Mediprobe Research Inc, London, Ontario
  - SKDS Research Inc, Newmarket, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Office of Dr. Michael Robern, Ottawa, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - K Papp Clinical Research Inc, Waterloo, Ontario
  - Recherche GCP Research, Montreal, Quebec
  - Dr. David Gratton Dermatologue Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain (CRDQ), Ste-Foy, Quebec
- Czechia (8):
  - CCBR Czech Prague s.r.o, Prague, Czech Republic
  - Dermatologie - MUDr. HELENA KORANDOVA s.r.o., Olomouc, Povel
  - CCBR Czech Brno, s.r.o, Brno
  - CCBR Czech a.s, Pardubice
  - Clintrial s.r.o, Prague
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - MUDr. Jaroslav Dragon - Kozni ordinace, Ústí nad Labem
  - Krajska zdravotni a.s. - Masarykova nemocnice v Usti nad Labem Dermatovenerologicke oddeleni, Ústí nad Labem
- Estonia (7):
  - Parnu Hospital, Pärnu
  - Vahlberg & Pild OU, Tallinn
  - East Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Medicum AS, Tallinn
  - Kliiniliste Uuringute Keskus (Clinical Research Centre), Tartu
  - Tartu University Hospital; Dermatology Clinic, Tartu
- Germany (6):
  - Universitaetsklinikum Schleswig Holstein, Schleswig, Holstein
  - Klinische Forschunq Schwerin GmbH, Dorf Mecklenburg, Vorpommern
  - Praxis fuer Dermatologie und Venerologie, Dresden
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main
  - Clinical Research Hamburg, Hamburg
- Latvia (5):
  - Riga 1 st Hospital, Riga
  - Derma Clinic Riga Ltd, Riga
  - Health Centre 4, Riga
  - J. Kisis Ltd, Riga
  - Ventspils Outpatient Clinic, Ventspils
- Poland (19):
  - Medica Pro Familia Sp. z o.o. S.K.A., Warsaw, Masovian Voivodeship
  - Poradnia Kardiologiczna Jaroslaw Jurowiecki, Gdansk
  - Medica Pro Familia Sp. z o. o. S.K.A. Oddzial w Gdyni, Gdynia
  - NZOZ POLIMEDICA FILIA KIELCE (Niepubliczny Zaklad Opieki Zdrowotnej POLIMEDICA), Kielce
  - Medica Pro Familia Sp. z o.o. SK.A., Krakow
  - Grazyna Pulka Specjalistyczny Osrodek ALL-MED, Krakow
  - Centrum Terapii Wspolczesnej _J.M. Jasnorzewska Sp. Komandytowo-Akcyjna, Lodz
  - Centrum Medyczne Szpital Swietej Rodziny, Lodz
  - NZOZ ALL-MED Centrum Medyczne Specjalistyczne Gabinety Lekarskie, Lodz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - Medicome sp.zoo, Oświęcim
  - Centrum Badan Klinicznych S.C., Poznan
  - Ai Centrum Medyczne, Poznan
  - KO-MED Centra Kliniczne Pulawy, Puławy
  - Centrum Medyczne Medyk, Rzeszów
  - NZOZ Nasz Lekarz, Torun
  - MTZ Clinical Research Sp z o.o., Warsaw
  - KO-MED Centra Kliniczne Zamosc, Zamość
  - Nzoz Polimedica, Zgierz
- Slovakia (5):
  - Pedi-Derma s.r.o., Košice, Košice Region
  - Derma therapy spol. s.r.o., Bratislava
  - Nemocnica Kosice-Saca, a.s., 1.sukromna nemocnica, Košice
  - Dema-beauty, s.r.o, Nitra
  - Sanare S.r.o, Svidník

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 572 participants were enrolled and randomized equally into M923 and European Union reference protein product (EU RPP) arms. One participant in each arm did not receive any treatment. The 263 participants completing EU RPP treatment in Part 1 were randomized to 1 of 2 treatment arms in Part 2 (Transition and Continuous).
Groups:
- Part 1 and Part 2: M923: Participants received 80 milligrams (mg) M923 (recombinant human immunoglobulin G subclass 1 [IgG1] monoclonal antibody specific for human tumor necrosis factor-alpha [TNF-α]) at Baseline (Week 0) and 40 mg every 2 weeks from Week 1 to Week 16 as a subcutaneous injection. Participants who received M923 in Part 1 continued to receive 40 mg M923 every 2 weeks from Week 17 to Week 48 (last dose at Week 47) as a subcutaneous injection.
- Part 1: EU RPP: Participants received 80 mg European Union Reference Protein Product (EU RPP) at Baseline (Week 0) and 40 mg every 2 weeks from Week 1 to Week 16 as a subcutaneous injection
- Part 1: EU RPP; Part 2: Transition: Participants received 80 mg EU RPP at Baseline (Week 0) and 40 mg every 2 weeks from Week 1 to Week 16 as a subcutaneous injection. At Week 17, participants who received EU RPP in Part 1 transitioned from EU RPP to M923 (40 mg every 2 weeks), then to EU RPP at Week 25 (40 mg every 2 weeks), and then to M923 at Week 37 (last dose at Week 47).
- Part 1: EU RPP; Part 2: Continous: Participants received 80 mg EU RPP at Baseline (Week 0) and 40 mg every 2 weeks from Week 1 to Week 16 as a subcutaneous injection. Participants who received EU RPP in Part 1 continued to receive EU RPP (40 mg every 2 weeks) from Week 17 to Week 48 (last dose at Week 47).
Period: Part 1: up to Week 16
Arm/Group | Part 1 and Part 2: M923 | Part 1: EU RPP | Part 1: EU RPP; Part 2: Transition | Part 1: EU RPP; Part 2: Continous
Started | 286 | 286 | 0 | 0
Completed | 271 | 263 | 0 | 0
Not Completed | 15 | 23 | 0 | 0
Not completed — Adverse Event | 3 | 8 | 0 | 0
Not completed — Physician Decision | 2 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 7 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Unspecified Reason | 3 | 3 | 0 | 0
Not completed — Did Not Receive Treatment | 1 | 1 | 0 | 0
Period: Part 2: Week 17 to Week 47
Arm/Group | Part 1 and Part 2: M923 | Part 1: EU RPP | Part 1: EU RPP; Part 2: Transition | Part 1: EU RPP; Part 2: Continous
Started | 271 | 0 | 132 | 131
Completed | 242 | 0 | 117 | 119
Not Completed | 29 | 0 | 15 | 12
Not completed — Adverse Event | 5 | 0 | 2 | 2
Not completed — Physician Decision | 3 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 9 | 0 | 7 | 5
Not completed — Failure to Achieve at Least a PASI 50 | 8 | 0 | 3 | 2
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1
Not completed — Unspecified Reason | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Analysis Set: all consenting participants randomized to study treatment
Groups:
- Part 1 and Part 2: M923: Participants received 80 milligrams (mg) M923 (recombinant human immunoglobulin G subclass 1 [IgG1] monoclonal antibody specific for human tumor necrosis factor-alpha [TNF-α]) at Baseline (Week 0) and 40 mg every 2 weeks from Week 1 to Week 48 as a subcutaneous injection.
- Part 1 and Part 2: EU RPP: Participants received 80 mg European Union Reference Protein Product (EU RPP) at Baseline (Week 0) and 40 mg every 2 weeks from Week 1 to Week 16 as a subcutaneous injection. Participants from this arm were then randomized at Week 16 into either Arm: Continuous EU RPP (continued EU RPP from Weeks 17 to 48 [last dose at Week 47]) or Arm: Transition EU RPP (transition to M923 at Week 17; then to EU RPP at Week 25; and then to M923 at Week 37 [last dose at Week 47]).
- Total: Total of all reporting groups
Arm/Group | Part 1 and Part 2: M923 | Part 1 and Part 2: EU RPP | Total
Number analyzed (Participants) | 286 | 286 | 572
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (12.4) | 45.5 (12.9) | 45.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 100 | 195
  Male | 191 | 186 | 377
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 281 | 282 | 563
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Psoriasis Area and Severity Index (PASI) Score [Mean (Standard Deviation); unit: units on a scale] — The PASI measures the average redness (erythema), thickness (induration), and scaliness [each graded on a scale of 0 (no disease) to 4 (very severe)] of psoriasis lesions, weighted by the area of involvement. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease. Population: Analysis was conducted using the Modified Intent-to-treat (mITT) Analysis Set including all consenting subjects randomized to study treatment (Arm A or Arm B) and contributed post-baseline data for at least one efficacy endpoint.
  units on a scale
    number analyzed (Participants) | 285 | 285 | 570
    (all) | 21.24 (9.27) | 20.16 (8.16) | 20.70 (8.74)
Number of Participants with the Indicated Static Physician's Global Assessment (sPGA) Score [Count of Participants; unit: Participants] — The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema). Population: mITT Analysis Set
  Participants
    number analyzed (Participants) | 285 | 285 | 570
    Moderate | 170 | 182 | 352
    Severe | 103 | 91 | 194
    Very Severe | 12 | 12 | 24
    Clear | 0 | 0 | 0
    Almost Clear | 0 | 0 | 0
    Mild | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a 75% Reduction in Psoriasis Area and Severity Index (PASI) (PASI 75) Scores at Week 16
Description: The PASI combines assessments of the extent of body surface involvement in 4 anatomical regions (head, arms, trunk, and legs) and the severity of scaling, redness, and thickness in each region, yielding an overall score of 0 for no disease to 72 for the most severe disease. Each of the body areas was scored by itself, and then the 4 scores were combined into the final PASI score. Participants achieving PASI 75 are defined as having an improvement (reduction) of at least 75% in the Week 16 PASI score compared to the score at Baseline.
Time Frame: Baseline; Week 16
Population: Per Protocol (PP) Analysis Set: subgroup of the Intent-To-Treat (ITT) Analysis Set that included all participants who did not have any deviations from the protocol deemed significant enough for exclusion from the efficacy analysis and received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 1: M923: Participants received 80 milligrams (mg) M923 (recombinant human immunoglobulin G subclass 1 [IgG1] monoclonal antibody specific for human tumor necrosis factor-alpha [TNF-α]) at Baseline (Week 0) and 40 mg every 2 weeks from Week 1 to Week 16 as a subcutaneous injection.
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 267 | 271
percentage of participants | 80.1 [74.9 to 84.8] | 79.0 [73.6 to 83.7]
Statistical Analysis 1: Comparison: Part 1: M923 vs Part 1: EU RPP; Test type: Equivalence — Per Food and Drug Administration (FDA), the equivalence testing was made using 90% confidence interval and an equivalence margin of 18%; Difference in proportion (M923 - EU RPP) = 0.014, 90% CI 2-sided [-0.043 to 0.072]
Statistical Analysis 2: Comparison: Part 1: M923 vs Part 1: EU RPP; Test type: Equivalence — Per European Medicines Agency (EMA), the equivalence testing was made using 95% confidence interval and an equivalence margin of 15%; Difference in proportion (M923 - EU RPP) = 0.014, 95% CI 2-sided [-0.054 to 0.082]

2. Secondary Outcome: Percentage of Participants With a Response of Clear or Almost Clear on the Static Physician Global Assessment (sPGA) at Week 16
Description: The sPGA response rate was defined as the percentage of participants who had achieved a clear or almost clear response on the 6-point sPGA scale. The sPGA was the physician's determination of the participant's psoriasis lesions overall at a given time point. Overall lesions were categorized by descriptions for induration, erythema, and scaling. For the analysis of responses, the participant's psoriasis was assessed at a given time point on a 6-point scale on which 0 = cleared, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, and 5 = very severe.
Time Frame: Week 16
Population: PP Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 1: M923: Participants received 80 mg M923 at Baseline (Week 0) and 40 mg every 2 weeks from Week 1 to Week 16 as a subcutaneous injection.
- Part 1: EU RPP: Participants received 80 mg EU RPP at Baseline (Week 0) and 40 mg every 2 weeks from Week 1 to Week 16 as a subcutaneous injection.
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 267 | 271
percentage of participants | 68.9 [63.0 to 74.4] | 66.1 [60.1 to 71.7]
Statistical Analysis 1: Comparison: Part 1: M923 vs Part 1: EU RPP; Test type: Other — No formal hypothesis testing of equivalence was performed for the comparison between M923 and EU RPP using the secondary efficacy outcome measures. Confidence Interval for difference in proportion in original scale was calculated using stratified Newcombe method; Difference in proportion (M923 - EU RPP) = 0.031, 95% CI 2-sided [-0.048 to 0.110]

3. Secondary Outcome: Number of Participants Achieving PASI 50 Response at Week 16
Description: The PASI combines assessments of the extent of body surface involvement in 4 anatomical regions (head, arms, trunk, and legs) and the severity of scaling, redness, and thickness in each region, yielding an overall score of 0 for no disease to 72 for the most severe disease. Each of the body areas was scored by itself, and then the 4 scores were combined into the final PASI score. Participants achieving PASI 50 are defined as having an improvement (reduction) of at least 50% compared to Baseline.
Time Frame: Baseline; Week 16
Population: PP Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 267 | 271
Participants | 243 | 253
Statistical Analysis 1: Comparison: Part 1: M923 vs Part 1: EU RPP; Test type: Other — No formal hypothesis testing of equivalence was performed for the comparison between M923 and EU RPP using the secondary efficacy outcome measures. Confidence Interval for difference in proportion in original scale calculated using stratified Newcombe method. Protocol defined margins are: [-0.18;+0.18] for 90% confidence interval; Difference in proportion (M923 - EU RPP) = -0.022, 90% CI 2-sided [-0.061 to 0.016]
Statistical Analysis 2: Comparison: Part 1: M923 vs Part 1: EU RPP; Test type: Other — No formal hypothesis testing of equivalence was performed for the comparison between M923 and EU RPP using the secondary efficacy outcome measures. Confidence Interval for difference in proportion in original scale calculated using stratified Newcombe method. Protocol defined margins are: [-0.15;+0.15] for 95% confidence interval; Difference in proportion (M923 - EU RPP) = -0.022, 95% CI 2-sided [-0.069 to 0.024]

4. Secondary Outcome: Number of Participants Achieving PASI 50 Response at Week 52 (Follow-Up Visit)
Description: as for outcome 3
Time Frame: Baseline; Week 52
Population: PP Analysis Set. Only those participants contributing data at Week 52 were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: M923: Participants who received M923 in Part 1 continued to receive 40 mg M923 every 2 weeks from Week 17 to Week 48 (last dose at Week 47) as a subcutaneous injection.
- Part 2: Transition EU RPP: At Week 17, participants who received EU RPP in Part 1 transitioned from EU RPP to M923 (40 mg every 2 weeks), then to EU RPP at Week 25 (40 mg every 2 weeks), and then to M923 at Week 37 (last dose at Week 47).
- Part 2: Continuous EU RPP: Participants who received EU RPP in Part 1 continued to receive EU RPP (40 mg every 2 weeks) from Week 17 to Week 48 (last dose at Week 47).
Arm/Group | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 258 | 130 | 129
Participants | 228 | 111 | 113

5. Secondary Outcome: Number of Participants Achieving PASI 75 Response at Week 52 (Follow-Up Visit)
Description: The PASI combines assessments of the extent of body surface involvement in 4 anatomical regions (head, arms, trunk, and legs) and the severity of scaling, redness, and thickness in each region, yielding an overall score of 0 for no disease to 72 for the most severe disease. Each of the body areas was scored by itself, and then the 4 scores were combined into the final PASI score. Participants achieving PASI 75 are defined as having an improvement (reduction) of at least 75% compared to Baseline.
Time Frame: Baseline; Week 52
Population: PP Analysis Set. Only those participants contributing data at Week 52 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 258 | 130 | 129
Participants | 202 | 96 | 101

6. Secondary Outcome: Number of Participants Achieving PASI 90 Response at Week 16
Description: The PASI combines assessments of the extent of body surface involvement in 4 anatomical regions (head, arms, trunk, and legs) and the severity of scaling, redness, and thickness in each region, yielding an overall score of 0 for no disease to 72 for the most severe disease. Each of the body areas was scored by itself, and then the 4 scores were combined into the final PASI score. Participants achieving PASI 90 are defined as having an improvement (reduction) of at least 90% compared to Baseline.
Time Frame: Baseline; Week 16
Population: PP Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 267 | 271
Participants | 165 | 147
Statistical Analysis 1: Comparison: Part 1: M923 vs Part 1: EU RPP; Test type: Other — [test comment as in outcome 3, analysis 1]; Difference in proportion (M923 - EU RPP) = 0.080, 90% CI 2-sided [0.010 to 0.149]
Statistical Analysis 2: Comparison: Part 1: M923 vs Part 1: EU RPP; Test type: Other — No formal hypothesis testing of equivalence was performed for the comparison between M923 and EU RPP using the secondary efficacy outcome measures. Confidence Interval for difference in proportion in original scale calculated using stratified Newcombe method. Protocol defined margins are:[-0.15;+0.15] for 95% confidence interval; Difference in proportion (M923 - EU RPP) = 0.080, 95% CI 2-sided [-0.004 to 0.162]

7. Secondary Outcome: Number of Participants Achieving PASI 90 Response at Week 52 (Follow-Up Visit)
Description: as for outcome 6
Time Frame: Baseline; Week 52
Population: PP Analysis Set. Only those participants contributing data at Week 52 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 258 | 130 | 129
Participants | 159 | 71 | 77

8. Secondary Outcome: Absolute PASI Score at Baseline
Description: The PASI combines assessments of the extent of body surface involvement in 4 anatomical regions (head, arms, trunk, and legs) and the severity of scaling, redness, and thickness in each region, yielding an overall score of 0 for no disease to 72 for the most severe disease. Each of the body areas was scored by itself, and then the 4 scores were combined into the final PASI score.
Time Frame: Baseline
Population: Analysis was performed using PP Analysis Set including participants with evaluable data for part 1 and part 2 of the study are included in the analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 267 | 271
units on a scale | 21.34 (9.268) | 20.29 (8.266)

9. Secondary Outcome: Absolute PASI Score at Week 16
Description: as for outcome 8
Time Frame: Week 16
Population: PP Analysis Set. Only those participants contributing data at Week 16 were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 261 | 263
units on a scale | 2.58 (4.092) | 2.50 (3.098)

10. Secondary Outcome: Absolute PASI Score at Week 52 (Follow-Up Visit)
Description: as for outcome 8
Time Frame: Week 52
Population: PP Analysis Set. Only those participants contributing data at Week 52 were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 246 | 120 | 124
units on a scale | 2.76 (4.768) | 2.85 (4.913) | 2.67 (3.919)

11. Secondary Outcome: Percent Change From Baseline in PASI Score at Week 16
Description: The PASI combines assessments of the extent of body surface involvement in 4 anatomical regions (head, arms, trunk, and legs) and the severity of scaling, redness, and thickness in each region, yielding an overall score of 0 for no disease to 72 for the most severe disease. Each of the body areas was scored by itself, and then the 4 scores were combined into the final PASI score. Percent change from Baseline was calculated as: (post-Baseline value - Baseline value) / (Baseline value) * 100.
Time Frame: Baseline; Week 16
Population: PP Analysis Set. Only those participants contributing data at Week 16 were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 261 | 263
percent change | -86.21 (20.065) | -86.79 (15.756)

12. Secondary Outcome: Percent Change From Baseline in PASI Score at Week 52 (Follow-Up Visit)
Description: as for outcome 11
Time Frame: Baseline; Week 52
Population: PP Analysis Set. Only those participants contributing data at Week 52 were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 246 | 120 | 124
percent change | -86.43 (22.570) | -85.53 (21.771) | -85.64 (20.968)

13. Secondary Outcome: Health-Related Quality of Life During Treatment: Dermatology Life Quality Index (DLQI) Score at Baseline
Description: The DLQI score was calculated by summing the individual scores of each question at a given time point, resulting in a maximum score of 30 and a minimum score of 0. The higher the score, the more quality of life is impaired. For the analysis of responses, the participant's results were assessed on a scoring scale on which 3 = very much or yes (applicable to question 7 only), 2 = a lot, 1 = a little, 0 = not at all or not relevant. Interpretation of DLQI scoring can be taken as 0 - 1 = no effect at all on participant's life, 2 - 5 = small effect on participant's life, 6 - 10 = moderate effect on participant's life, 11 - 20 = very large effect on participant's life, and 21 - 30 = extremely large effect on participant's life.
Time Frame: Baseline
Population: Analysis was performed using PP Analysis Set including participants with evaluable data for part 1 and part 2 of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 267 | 271
units on a scale | 12.5 (7.13) | 10.5 (6.71)

14. Secondary Outcome: Health-Related Quality of Life During Treatment: DLQI Score at Week 16
Description: as for outcome 13
Time Frame: Week 16
Population: PP Analysis Set. Only those participants contributing data at Week 16 were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 258 | 259
units on a scale | 2.4 (4.04) | 2.1 (3.50)

15. Secondary Outcome: Health-Related Quality of Life During Treatment: DLQI Score at Week 48 (Completion/Termination Visit)
Description: as for outcome 13
Time Frame: Week 48
Population: PP Analysis Set. Only those participants contributing data at Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 232 | 115 | 117
units on a scale | 2.1 (3.77) | 1.6 (2.83) | 2.1 (3.97)

16. Secondary Outcome: Health-Related Quality of Life During Treatment: EuroQoL 5-Dimension Health Status Questionnaire (EQ-5D-5L) at Baseline
Description: The EQ-5D-5L health score was measured on a Visual Analog Scale (VAS) anchored by 0 = "worst health you can imagine" and 100 = "best health you can imagine". Baseline was defined as the last scheduled observation prior to dosing, typically Day 1, predose.
Time Frame: Baseline
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 267 | 271
units on a scale | 71.3 (18.70) | 72.5 (20.27)

17. Secondary Outcome: Health-Related Quality of Life During Treatment: EQ-5D-5L at Week 16
Description: The EQ-5D-5L health score was measured on a Visual Analog Scale (VAS) anchored by 0 = "worst health you can imagine" and 100 = "best health you can imagine".
Time Frame: Week 16
Population: PP Analysis Set. Only those participants contributing data at Week 16 were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 258 | 259
units on a scale | 83.7 (12.38) | 83.4 (13.92)

18. Secondary Outcome: Health-Related Quality of Life During Treatment: EQ-5D-5L at Week 48 (Completion/Termination Visit)
Description: as for outcome 17
Time Frame: Week 48
Population: PP Analysis Set. Only those participants contributing data at Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 232 | 115 | 117
units on a scale | 85.3 (13.83) | 83.9 (14.92) | 84.2 (12.98)

19. Secondary Outcome: Number of Participants With Clinically Meaningful Changes in Vital Signs
Description: Vital signs included body temperature, respiratory rate, pulse rate, systolic and diastolic blood pressure, and weight. Clinically meaningful changes were classified as such by the Investigator and reported as adverse events.
Time Frame: Up to Week 52
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: M923 | Part 1: EU RPP | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 285 | 285 | 271 | 132 | 131
Participants | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters at Baseline
Description: Laboratory results included hematology [Hemoglobin, Hematocrit, Platelet count, Mean cell volume, White blood cell count (total leucocytes), Neutrophils absolute, Neutrophils, Lymphocytes absolute, Lymphocytes, Monocytes, Eosinophils absolute, and Eosinophils], chemistry (Aspartate transaminase, Alanine transaminase, Gamma glutamyl transferase, Creatine kinase, C-reactive protein, Cholesterol, Triglycerides, Total protein, Potassium, Urea, Creatinine, Phosphate, Glucose, and Uric acid) and urinalysis [Specific Gravity] parameters. Laboratory results of a few hematology (Red Blood Cell Count and Monocytes absolute), chemistry (Alkaline Phosphatase, Total bilirubin, Sodium, Chloride, and Albumin), and urinalysis (pH) parameters were not assessed at Baseline and Week 16. Clinically meaningful changes were classified as such by the Investigator and reported as adverse events.
Time Frame: Baseline
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 285 | 285
Participants
  Hemoglobin | 0 | 0
  Hematocrit | 0 | 0
  Platelet count | 0 | 0
  Mean cell volume | 0 | 0
  White blood cell count (total leucocytes) | 1 | 1
  Neutrophils absolute | 2 | 1
  Neutrophils | 1 | 0
  Lymphocytes absolute | 1 | 1
  Lymphocytes | 1 | 1
  Monocytes | 0 | 0
  Eosinophils absolute | 0 | 0
  Eosinophils | 0 | 0
  Aspartate transaminase | 0 | 0
  Alanine transaminase | 1 | 1
  Gamma glutamyl transferase | 1 | 4
  Creatine kinase | 2 | 0
  C-reactive protein | 6 | 2
  Cholesterol | 2 | 4
  Triglycerides | 3 | 2
  Total protein | 0 | 1
  Potassium | 1 | 0
  Urea | 1 | 0
  Creatinine | 0 | 0
  Phosphate | 0 | 0
  Glucose | 1 | 2
  Uric acid | 2 | 0
  Specific Gravity | 0 | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters at Week 16
Description: as for outcome 20
Time Frame: Week 16
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 285 | 285
Participants
  Hemoglobin | 1 | 1
  Hematocrit | 1 | 1
  Platelet count | 0 | 0
  Mean cell volume | 0 | 1
  White blood cell count (total leucocytes) | 2 | 0
  Neutrophils absolute | 1 | 0
  Neutrophils | 0 | 0
  Lymphocytes absolute | 0 | 1
  Lymphocytes | 0 | 1
  Monocytes | 0 | 0
  Eosinophils absolute | 1 | 0
  Eosinophils | 1 | 0
  Aspartate transaminase | 2 | 0
  Alanine transaminase | 3 | 1
  Gamma glutamyl transferase | 3 | 2
  Creatine kinase | 2 | 0
  C-reactive protein | 1 | 0
  Cholesterol | 4 | 3
  Triglycerides | 5 | 3
  Total protein | 0 | 1
  Potassium | 1 | 0
  Urea | 0 | 0
  Creatinine | 0 | 0
  Phosphate | 0 | 0
  Glucose | 2 | 3
  Uric acid | 1 | 1
  Specific Gravity | 0 | 0

22. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters at Week 48 (Completion/Termination Visit)
Description: Laboratory results included hematology [Red Blood Cell Count, Hemoglobin, Hematocrit, Platelet count, Mean cell volume, White blood cell count (total leucocytes), Neutrophils absolute, Neutrophils, Lymphocytes absolute, Lymphocytes, Monocytes absolute, Monocytes, Eosinophils absolute, and Eosinophils], chemistry (Aspartate transaminase, Alanine transaminase, Alkaline Phosphatase, Gamma glutamyl transferase, Total bilirubin, Creatine kinase, C-reactive protein, Cholesterol, Triglycerides, Total protein, Sodium, Potassium, Chloride, Urea, Creatinine, Albumin, Phosphate, Glucose, and Uric acid) and urinalysis [pH and Specific Gravity] parameters. Clinically meaningful changes were classified as such by the Investigator and reported as adverse events.
Time Frame: Week 48
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 271 | 132 | 131
Participants
  Red Blood Cell Count | 1 | 0 | 1
  Hemoglobin | 1 | 0 | 1
  Hematocrit | 1 | 0 | 1
  Platelet count | 1 | 0 | 0
  Mean cell volume | 0 | 0 | 1
  White blood cell count (total leucocytes) | 2 | 1 | 1
  Neutrophils absolute | 3 | 1 | 2
  Neutrophils | 3 | 0 | 0
  Lymphocytes absolute | 0 | 0 | 1
  Lymphocytes | 1 | 0 | 0
  Monocytes absolute | 0 | 0 | 0
  Monocytes | 1 | 0 | 0
  Eosinophils absolute | 0 | 0 | 0
  Eosinophils | 2 | 0 | 0
  Aspartate transaminase | 2 | 0 | 1
  Alanine transaminase | 5 | 0 | 3
  Alkaline Phosphatase | 0 | 0 | 0
  Gamma glutamyl transferase | 3 | 0 | 3
  Total bilirubin | 1 | 0 | 1
  Creatine kinase | 0 | 1 | 1
  C-reactive protein | 3 | 0 | 0
  Cholesterol | 7 | 3 | 2
  Triglycerides | 11 | 4 | 2
  Total protein | 0 | 0 | 0
  Sodium | 0 | 0 | 0
  Potassium | 0 | 0 | 0
  Chloride | 0 | 0 | 0
  Urea | 0 | 0 | 0
  Creatinine | 0 | 0 | 0
  Albumin | 0 | 0 | 0
  Phosphate | 0 | 0 | 0
  Glucose | 5 | 3 | 0
  Uric acid | 1 | 3 | 3
  pH | 1 | 1 | 0
  Specific Gravity | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram Parameters at Baseline
Description: Clinically significant abnormalities were classified as such by the Investigator and reported as adverse events.
Time Frame: Baseline
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 285 | 285
Participants | 0 | 0

24. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram Parameters at Week 16
Description: Clinically significant abnormalities were classified as such by the Investigator and reported as adverse events.
Time Frame: Week 16
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 285 | 285
Participants | 2 | 0

25. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram Parameters at Week 48 (Completion/Termination Visit)
Description: Clinically significant abnormalities were classified as such by the Investigator and reported as adverse events.
Time Frame: Week 48
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 271 | 132 | 131
Participants | 3 | 0 | 0

26. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs are adverse events that occurred during or after study drug administration. For more details on adverse events please refer the safety section.
Time Frame: Up to Week 52
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: M923 | Part 1: EU RPP | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 285 | 285 | 271 | 132 | 131
Participants | 169 | 194 | 199 | 99 | 103

27. Secondary Outcome: Pharmacokinetics: Serum Concentrations by Treatment
Description: Serum samples were collected at Baseline (Week 0, perdose), approximately 1 week (peak) after IP administration (Weeks 8 and 16), and 2 weeks after dose administration as a trough sample collected prior to the next dose administration (Weeks 17, 21, 25, 29, 37, 41).
Time Frame: Baseline (Week 0), Week 8, 16, 17, 21, 25, 29, 37, and 41
Population: Pharmacokinetic (PK) Analysis Set: all participants who received at least 1 dose of study drug and had at least 1 measured concentration at a scheduled PK time point after start of dosing. Only participants with evaluable data were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliter (ng/mL)
Arm/Group | Part 1: M923 | Part 1: EU RPP | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 282 | 281 | 267 | 130 | 130
nanograms per milliter (ng/mL)
  Baseline (Week 0)/Predose: number analyzed (Participants) | 279 | 279 | 0 | 0 | 0
  Baseline (Week 0)/Predose | 302 (16.5) | 301 (9.69) |  |  |
  Week 8/Peak: number analyzed (Participants) | 277 | 272 | 0 | 0 | 0
  Week 8/Peak | 9100 (5450) | 7640 (4370) |  |  |
  Week 16/Peak: number analyzed (Participants) | 268 | 261 | 0 | 0 | 0
  Week 16/Peak | 8580 (5700) | 6990 (5100) |  |  |
  Week 17/Trough: number analyzed (Participants) | 0 | 0 | 267 | 130 | 129
  Week 17/Trough |  |  | 6900 (5270) | 5840 (4840) | 5340 (4050)
  Week 21/Trough: number analyzed (Participants) | 0 | 0 | 257 | 127 | 130
  Week 21/Trough |  |  | 6630 (4960) | 6260 (4960) | 5100 (4040)
  Week 25/Trough: number analyzed (Participants) | 0 | 0 | 252 | 126 | 127
  Week 25/Trough |  |  | 6790 (5210) | 6320 (5260) | 4970 (3870)
  Week 29/Trough: number analyzed (Participants) | 0 | 0 | 248 | 125 | 124
  Week 29/Trough |  |  | 5990 (4020) | 5330 (4000) | 4840 (3480)
  Week 37/Trough: number analyzed (Participants) | 0 | 0 | 245 | 121 | 120
  Week 37/Trough |  |  | 6120 (4220) | 5250 (4190) | 4830 (3680)
  Week 41/Trough: number analyzed (Participants) | 0 | 0 | 241 | 119 | 117
  Week 41/Trough |  |  | 5950 (4230) | 5480 (4140) | 4740 (3710)

28. Secondary Outcome: Immunogenicity: Number of Participants With Anti-Drug Antibodies (ADA) at Baseline
Description: The M923 confirmation assay was evaluated only if the EU Humira confirmation assay was negative. Overall Result: a participant was considered to be positive if a confirmed positive result was observed at any assay (including predose; if a participant had either a negative result in the screening assay or a positive result at screening followed by a negative result in all confirmation tiers, the overall result was negative. Overall Status: a participant was considered to have developed ADA or neutralizing ADAs if a confirmed positive result was observed at any time during the treatment period inclusive of the predose results; the designation of negative required either a negative screening assay or a negative confirmation result at each sampling time. The same convention applied for the neutralizing assay results.
Time Frame: Baseline (Week 0)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 285 | 285
Participants
  EU Humera | 15 | 11
  M923 | 1 | 2
  Overall Results | 16 | 13
  Neutralizing ADA | 4 | 2

29. Secondary Outcome: Immunogenicity: Number of Participants With ADA at Week 16
Description: as for outcome 28
Time Frame: Week 16
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 285 | 285
Participants
  EU Humera | 135 | 144
  M923 | 4 | 8
  Overall Results | 139 | 152
  Neutralizing ADA | 28 | 30

30. Secondary Outcome: Immunogenicity: Number of Participants With ADA at Week 25
Description: as for outcome 28
Time Frame: Week 25
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 271 | 132 | 131
Participants
  EU Humera | 144 | 80 | 92
  M923 | 12 | 5 | 5
  Overall result | 156 | 85 | 97
  Neutralizing ADA | 55 | 25 | 32

31. Secondary Outcome: Immunogenicity: Number of Participants With ADA at Week 52 (Completion/Termination Visit)
Description: as for outcome 28
Time Frame: Week 52
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 271 | 132 | 131
Participants
  EU Humera | 131 | 73 | 80
  M923 | 10 | 6 | 7
  Overall result | 141 | 79 | 87
  Neutralizing ADA | 40 | 28 | 23

32. Secondary Outcome: Immunogenicity: Number of Participants With ADA and nADA by Titer at Baseline
Description: The M923 confirmation assay was evaluated only if the EU Humira confirmation assay was negative. Overall Result: a participant was considered to be positive if a confirmed positive result was observed at any assay (including predose); if a participant had either a negative result in the screening assay or a positive result at screening followed by a negative result in all confirmation tiers, the overall result was negative. Overall Status: a participant was considered to have developed ADA or neutralizing ADAs if a confirmed positive result was observed at any time during the treatment period inclusive of the predose results; the designation of negative required either a negative screening assay or a negative confirmation result at each sampling time. In confirmed positive samples, an assay was used to determine the relative titer of the ADA; a subsequent neutralizing antibodies assay was used to determine the presence of neutralizing antibodies.
Time Frame: Baseline (Week 0)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 285 | 285
Participants
  No positive result | 266 | 271
  Predose positive result | 16 | 13

33. Secondary Outcome: Immunogenicity: Number of Participants With ADA and nADA by Titer at Week 16
Description: as for outcome 32
Time Frame: Week 16
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: M923 | Part 1: EU RPP
Number analyzed (Participants) | 285 | 285
Participants
  Titers ≤ 1:16 (postdose positive ADAs) | 16 | 26
  Titers ≤ 1:16 (postdose positive nADAs) | 2 | 2
  Titers > 1:16 to ≤ 1:128 (postdose positive ADAs) | 90 | 73
  Titers > 1:16 to ≤ 1:128 (postdose positive nADAs) | 17 | 6
  Titers >1:128 to ≤ 1:152 (postdose positive ADAs) | 27 | 40
  Titers >1:128 to ≤ 1:152 (postdose positive nADAs) | 3 | 11
  Titers >1:152 (postdose positive ADAs) | 6 | 13
  Titers >1:152 (postdose positive nADAs) | 6 | 11

34. Secondary Outcome: Immunogenicity: Number of Participants With ADA and nADA by Titer at Week 25
Description: as for outcome 32
Time Frame: Week 25
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 and Part 2: M923: Participants received 80 mg M923 at Baseline (Week 0) and 40 mg every 2 weeks from Week 1 to Week 48 as a subcutaneous injection.
Arm/Group | Part 1 and Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 285 | 132 | 131
Participants
  Titers ≤ 1:16 (postdose positive ADAs) | 24 | 19 | 21
  Titers ≤ 1:16 (postdose positive nADAs) | 6 | 2 | 4
  Titers > 1:16 to ≤ 1:128 (postdose positive ADAs) | 86 | 37 | 42
  Titers > 1:16 to ≤ 1:128 (postdose positive nADAs) | 17 | 4 | 7
  Titers >1:128 to ≤ 1:152 (postdose positive ADAs) | 28 | 14 | 22
  Titers >1:128 to ≤ 1:152 (postdose positive nADAs) | 16 | 6 | 10
  Titers >1:152 (postdose positive ADAs) | 18 | 15 | 12
  Titers >1:152 (postdose positive nADAs) | 16 | 13 | 11

35. Secondary Outcome: Immunogenicity: Number of Participants With ADA and nADA by Titer at Week 52 (Completion/Termination Visit)
Description: as for outcome 32
Time Frame: Week 52
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 and Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 285 | 132 | 131
Participants
  Titers ≤ 1:16 (postdose positive ADAs) | 26 | 11 | 17
  Titers ≤ 1:16 (postdose positive nADAs) | 0 | 2 | 3
  Titers > 1:16 to ≤ 1:128 (postdose positive ADAs) | 62 | 37 | 38
  Titers > 1:16 to ≤ 1:128 (postdose positive nADAs) | 13 | 6 | 5
  Titers >1:128 to ≤ 1:152 (postdose positive ADAs) | 23 | 12 | 15
  Titers >1:128 to ≤ 1:152 (postdose positive nADAs) | 9 | 6 | 2
  Titers >1:152 (postdose positive ADAs) | 13 | 7 | 10
  Titers >1:152 (postdose positive nADAs) | 11 | 6 | 7

36. Secondary Outcome: Median Time to Seroconversion
Description: Time to seroconversion (in days) was defined as the time to the observation of the first confirmed positive ADA response. Participants with confirmed positive ADA response at baseline (Week 0 predose) were excluded.
Time Frame: Up to Week 52
Population: Safety Analysis Set. Only those participants who had a postdose seroconversion time were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Part 1 and Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
Number analyzed (Participants) | 216 | 106 | 120
days | 113.0 [52 to 372] | 113.0 [51 to 375] | 112.0 [54 to 373]

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: Adverse events were collected in members of the Safety Analysis Set, comprised of all participants who received at least 1 dose of study drug (M923 or European Union reference protein product [EU RPP]).
Arm/Group | Part 1: M923 | Part 1: EU RPP | Part 2: M923 | Part 2: Transition EU RPP | Part 2: Continuous EU RPP
All-Cause Mortality (participants affected / at risk) | 0/285 | 0/285 | 0/271 | 0/132 | 0/131
Serious Adverse Events (participants affected / at risk) | 4/285 | 7/285 | 10/271 | 10/132 | 8/131
Other Adverse Events (participants affected / at risk) | 92/285 | 104/285 | 96/271 | 47/132 | 63/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: M923 (N=285) | Part 1: EU RPP (N=285) | Part 2: M923 (N=271) | Part 2: Transition EU RPP (N=132) | Part 2: Continuous EU RPP (N=131)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Benign ovarian tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Device loosening (Product Issues) | 0 | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Genital prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: M923 (N=285) | Part 1: EU RPP (N=285) | Part 2: M923 (N=271) | Part 2: Transition EU RPP (N=132) | Part 2: Continuous EU RPP (N=131)
Injection site reaction (General disorders) | 68 | 79 | 27 | 15 | 19
Nasopharyngitis (Infections and infestations) | 19 | 17 | 40 | 16 | 20
Upper respiratory tract infection (Infections and infestations) | 9 | 6 | 15 | 6 | 11
Headache (Nervous system disorders) | 9 | 10 | 2 | 7 | 5
Psoriasis (Skin and subcutaneous tissue disorders) | 8 | 8 | 28 | 14 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT02581345/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT02581345/SAP_001.pdf